CLINICAL TRIAL: NCT07052448
Title: The Efficacy of Sequential Radiotherapy After the Combination of Transcatheter Arterial Chemoembolization With Lenvatinib and Anti-PD-1 Antibodies for Unresectable Hepatocellular Carcinoma
Brief Title: The Efficacy of Sequential RT After Triple Therapy for uHCC
Status: Enrolling by invitation | Type: Observational
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Mao-Lin Yan, professor, Fujian Provincial Hospital
Other Study IDs: TALENP006
Record Dates: First submitted 2025-06-21; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- sequential radiotherapy after triple therapy: Patients with unresectable hepatocellular carcinoma received sequential radiotherapy after the combination of transcatheter arterial chemoembolization with lenvatinib and anti-PD-1 antibodies
  Interventions: Drug: sequential radiotherapy after the combination of transcatheter arterial chemoembolization (TACE) combined with lenvatinib and anti-PD-1 antibodies

INTERVENTIONS:
Drug: sequential radiotherapy after the combination of transcatheter arterial chemoembolization (TACE) combined with lenvatinib and anti-PD-1 antibodies — sequential radiotherapy after the combination of transcatheter arterial chemoembolization (TACE) combined with lenvatinib and anti-PD-1 antibodies

SUMMARY:
Triple therapy of transcatheter arterial chemoembolization (TACE) combined with lenvatinib and anti-PD-1 antibodies has demonstrated excellent efficacy in unresectable hepatocellular carcinoma (uHCC). However, tumor drug resistance is still a major problem and many patients fail to achieve complete necrosis of the lesions after treatment. This study aimed to investigate the efficacy and safety of sequential radiotherapy after triple therapy in patients with uHCC to improve tumor response rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with HCC and assessed as unresectable by multidisciplinary team (MDT)
* Patients who achieved PR or SD after triple therapy according to the mRECIST and did not meet the criteria for radical surgical resection or could not tolerate surgical treatment
* Patients who received sequential radiotherapy
* Age between 18 and 75 years
* Child-Pugh class A or B
* Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0-1

Exclusion Criteria:

* Previous acceptance of other antitumor treatments
* Treatment in conjunction with other treatment regimens, such as radiofrequency ablation and chemotherapy
* History of other malignancies
* Incomplete data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable hepatocellular carcinoma received sequential radiotherapy after the combination of transcatheter arterial chemoembolization with lenvatinib and anti-PD-1 antibodies.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
OS | From date of randomization until the date of date of death from any cause or the most recent follow-up, whichever came first, assessed up to 100 months
  overall survival

SECONDARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression, the date of death from any cause or the date of most recent follow-up, whichever came first, assessed up to 100 months
  progression-free survival
ORR | From date of randomization until the date of the best tumor response is achieved, assessed up to 100 months
  objective response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Fuzhou University Affiliated Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are not publicly available due to privacy reasons but are available from the corresponding author upon reasonable request.